CLINICAL TRIAL: NCT04652271
Title: PancreasGroup.Org - International Pancreatic Surgery Outcomes Study
Brief Title: International Pancreatic Surgery Outcomes Study - PancreasGroup.Org
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: University College London Hospitals (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20203109-PG
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Pancreatic Neoplasms; Pancreatitis
Keywords: pancreatic surgery; snapshot; global surgery; predictors; outcomes
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing pancreatic surgery: Patients undergoing any type of pancreatic surgery.
  Interventions: Procedure: Pancreatic surgery

INTERVENTIONS:
Procedure: Pancreatic surgery — Open, laparoscopic or robotic surgery of the pancreas

SUMMARY:
"Snapshot" study worldwide over 3 months in 2021. Provide a verified record of true morbidity and mortality. Identify modifiable predicting factors of outcome. Obtain PubMed citable co-authorship,

DETAILED DESCRIPTION:
The PancreasGroup.org team is conducting a "snapshot" clinical study investigating the outcomes of pancreatic surgery worldwide. This "collaborative" model for snapshot clinical studies is a well-established approach for assessing current practice in a short period of time.

There will be 3 months of prospective enrolment and 3 months follow up within a 12-month frame. The study will provide highly valuable data on outcomes after pancreatic surgery.

The investigators are aiming at providing a verified record of true morbidity and mortality in consecutive unselected patients. This way the investigators will help identify relevant, modifiable predicting factors for outcome after pancreatic surgery.

ELIGIBILITY:
Inclusion Criteria:

* All indications (including benign and malignant)
* Open, laparoscopic or robotic.
* Elective or emergency.
* Partial or total pancreatectomies.
* Pancreatic tumour enucleations.
* Procedures with concomitant vascular or other organ resections.
* Pancreatic duct drainage procedures (e.g. Frey, Puestow, or Beger)
* Adults 18 years of age or older.

Exclusion Criteria:

* Pancreas or islet cell transplantation.
* Transcutaneous or transgastric imaging-guided ablation (e.g. RFA) or electroporation (e.g. NanoKnife).
* Endoscopic (e.g. endoscopic retrograde cholangiopancreatography, stent or lithotripsy) procedures.
* Endoscopic transgastric and surgical necrosectomies excluded.
* Patients less than 18 years of age excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing pancreatic resection by surgeons at their respective centres are eligible for study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days postoperatively
  Postoperative death

SECONDARY OUTCOMES:
Morbidity | 90 days postoperatively
  Postoperative complication rates classified according to Clavien-Dindo

CONTACTS AND LOCATIONS:
Overall Officials: Guiseppe K Fusai, MD, MS, Study Chair — Royal Free Hospital London, UK; Cristina Ferrone, MD, Study Chair — Massachusetts General Hospital, Boston, USA; Dimitri A Raptis, MD, MSc, PhD, Principal Investigator — Royal Free Hospital London, UK

IPD SHARING:
Plan to Share IPD: Yes
PancreasGroup.org is a collaboration of all surgeons contributing data as equal partners. Each surgeon contributing data has access to analysis files of the entire database at any time point and the right to propose analyses and publish data as long as every surgeon contributing data are included as a group author in every publication and have an opportunity to review the data prior to submission. Each collaborator has access to their own data in a form of excel export file without requiring permission or approval by the PancreasGroup.org management committee.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will become available after the first and main publication of PancreasGroup.org. They will be available for at least 10 years.

REFERENCES:
- [Derived] PancreasGroup.org Collaborative. Pancreatic surgery outcomes: multicentre prospective snapshot study in 67 countries. Br J Surg. 2024 Jan 3;111(1):znad330. doi: 10.1093/bjs/znad330. PMID 38743040
- See also: The official website of PancreasGroup.org — https://pancreasgroup.org/
- See also: The R statistical package for analysis — https://rbiostatistics.com